CLINICAL TRIAL: NCT06942013
Title: Radiographic Assessment of Cortical Shell Technique For Horizontal Ridge Augmentation In The Anterior Mandible Using Full Digital Workflow Versus Free Hand Protocol: A Randomized Clinical Trial
Brief Title: Radiographic Assessment of Guided Cortical Shell Technique for Horizontal Ridge Augmentation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mayar Momen El Khawass, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cortical Shell Technique
Record Dates: First submitted 2025-03-16; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Horizontal Ridge Deficiency
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Type: Parallel, two arms, randomized controlled trial Allocation ratio: 1:1 Framework: Equivalence
Who Masked: Participant
Masking Description: This trial is considered a randomized single blind clinical trial due to the following:
  1. The participants will be blinded to the technique that will be used during the surgical procedure.
  2. The operator (M.E.) will not be blinded for both techniques during the surgical procedure as the two techniques are different.
  3. The outcome assessor (Dr. S.H.) cannot be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Full Digital Workflow (Experimental): Study Group (Computer-Guided Autogenous Cortical Shell Technique)
  Bone harvesting and fixation are done using patient-specific guides , chin harvesting guide and bone block fixation guide. Uses a 3D-printed, patient-specific surgical guide for precise bone harvesting and placement.
  Piezo drill cuts are guided to ensure accurate osteotomy and graft positioning. The labial cortical shell is fixated using pre-planned screw holes for better stability.
  Bone particulate grafting (autogenous + xenograft, 50:50) is packed into the defect.
  Enhances accuracy, reduces surgical time, and minimizes complications
  Interventions: Device: Computer-Guided Autogenous Cortical Shell Technique (Study Group)
- Free Hand Protocol (Active Comparator): Control Group (Free-Hand Autogenous Cortical Shell Technique)
  Bone harvesting and fixation are done manually, relying on the surgeon's experience.
  Osteotomy is performed free-hand, increasing the risk of inaccurate graft placement.
  The labial cortical shell is manually fixated, potentially leading to misalignment.
  Bone particulate grafting (autogenous + xenograft, 50:50) is used, similar to the study group.
  Higher risk of human error, longer surgical time, and greater variability in outcomes
  Interventions: Procedure: Free-Hand Autogenous Cortical Shell Technique (Control group)

INTERVENTIONS:
Device: Computer-Guided Autogenous Cortical Shell Technique (Study Group) — This study utilizes two patient-specific 3D-printed surgical guides to enhance precision in bone harvesting and fixation for horizontal ridge augmentation in the anterior mandible.
  Chin Harvesting Guide
  This tooth-supported guide is placed on the exposed mandibular symphysis to ensure accurate osteotomy cuts for harvesting a cortical bone shell.
  It directs piezo drill cuts (superior, inferior, and vertical) to minimize errors and prevent damage to vital structures.
  Bone Block Fixation Guide
  After harvesting, this guide helps in precise fixation of the cortical shell onto the recipient site.
  It includes pre-planned screw holes to ensure stable positioning of the graft and improve surgical accuracy.
  These guides enhance precision, reduce surgical time, and improve graft stability, making the computer-guided technique superior to the traditional free-hand method.
  Arms: Full Digital Workflow
Procedure: Free-Hand Autogenous Cortical Shell Technique (Control group) — In this group, horizontal ridge augmentation of the anterior mandible is performed using a free-hand technique without computer-guided assistance. Autogenous cortical bone is harvested from the mandibular symphysis using a conventional osteotomy performed manually. The harvested cortical shell is adapted and fixated at the recipient site using titanium mini screws, based on the surgeon's clinical judgment and intraoperative assessment. Bone particulate grafting using a 1:1 ratio of autogenous bone and xenograft material is packed into the defect to enhance volume stability. This approach may result in increased variability in graft positioning, longer surgical time, and higher dependence on surgeon experience.
  Arms: Free Hand Protocol

SUMMARY:
The protocol outlines a randomized clinical trial comparing two surgical techniques for horizontal ridge augmentation in the anterior mandible:

Computer-Guided Autogenous Cortical Shell Technique (using a patient-specific guide for precise placement).

Free-Hand Autogenous Cortical Shell Technique (traditional approach without a guiding template).

Key Points:

The study aims to determine which method provides better accuracy and bone volume stability.

Cone Beam CT scans (CBCT) will assess horizontal bone gain preoperatively and six months postoperatively.

The trial is conducted at Cairo University's Faculty of Dentistry. Participants: Patients with pure horizontal bone loss in the anterior mandible.

Outcomes:

Primary: Bone width gain in millimeters. Secondary: Accuracy of augmentation and surgical time.

Methodology:

The study group will use computer-designed surgical osteotomy guides to harvest and place bone grafts with improved precision.

The control group will rely on the conventional free-hand approach. Both groups will undergo bone grafting using autogenous cortical bone shells.

Data Collection & Analysis:

Participants will be randomized and blinded. Data will be analyzed using statistical methods to compare effectiveness.

DETAILED DESCRIPTION:
This randomized controlled trial evaluates the clinical effectiveness and surgical accuracy of a computer-guided versus a conventional free-hand approach for horizontal ridge augmentation in the anterior mandible using the autogenous cortical shell technique.

Participants presenting with horizontal alveolar bone deficiency in the anterior mandible are randomly assigned to one of two groups:

Study Group: A fully digital workflow is employed, including CBCT-based virtual planning and the use of 3D-printed, patient-specific stereolithographic guides for both bone harvesting and graft placement.

Control Group: The traditional free-hand technique is used without computer-guided assistance.

The study is designed to assess whether the digital, guided approach enhances horizontal bone gain, optimizes graft placement accuracy, reduces operative time, and lowers complication rates compared to the free-hand protocol.

The intervention involves preoperative 3D planning, surgical guide fabrication, and intraoperative bone harvesting and grafting. Both groups receive autogenous cortical bone blocks harvested from the mandibular symphysis and secured at the recipient site with mini screws. Bone particulate (autogenous + xenograft, 1:1 ratio) is used to augment volume.

Primary outcome is the amount of horizontal bone gain measured via CBCT superimposition at baseline and 6 months postoperatively. Secondary outcomes include surgical time, accuracy of graft placement, and incidence of postoperative complications such as pain, swelling, infection, dehiscence, or graft exposure.

This single-center, single-blinded equivalence trial uses a 1:1 randomization ratio. Ethical approval has been obtained, and participants provide informed consent prior to enrollment. The results are expected to inform surgical best practices and improve the predictability of mandibular ridge augmentation procedures.This randomized controlled trial evaluates the clinical effectiveness and surgical accuracy of a computer-guided versus a conventional free-hand approach for horizontal ridge augmentation in the anterior mandible using the autogenous cortical shell technique.

Participants presenting with horizontal alveolar bone deficiency in the anterior mandible are randomly assigned to one of two groups:

Study Group: A fully digital workflow is employed, including CBCT-based virtual planning and the use of 3D-printed, patient-specific stereolithographic guides for both bone harvesting and graft placement.

Control Group: The traditional free-hand technique is used without computer-guided assistance.

The study is designed to assess whether the digital, guided approach enhances horizontal bone gain, optimizes graft placement accuracy, reduces operative time, and lowers complication rates compared to the free-hand protocol.

The intervention involves preoperative 3D planning, surgical guide fabrication, and intraoperative bone harvesting and grafting. Both groups receive autogenous cortical bone blocks harvested from the mandibular symphysis and secured at the recipient site with mini screws. Bone particulate (autogenous + xenograft, 1:1 ratio) is used to augment volume.

Primary outcome is the amount of horizontal bone gain measured via CBCT superimposition at baseline and 6 months postoperatively. Secondary outcomes include accuracy of graft placement, and surgical time.

This single-center, single-blinded equivalence trial uses a 1:1 randomization ratio. Ethical approval has been obtained, and participants provide informed consent prior to enrollment. The results are expected to inform surgical best practices and improve the predictability of mandibular ridge augmentation procedures.

ELIGIBILITY:
Inclusion Criteria:

* • Anterior mandible with horizontal deficient alveolar ridge that is from 2 to 4 mm measured from the crest of the alveolar ridge buccolingually.

  * Class IV and V according to Cawood and Howell classification.
  * No sex predilection.
  * Patients free from any systemic conditions and bone metabolism diseases that might interfere with the surgical intervention, soft tissue or hard tissue healing.
  * The minimum number of missing teeth in the anterior mandible alveolar ridge is two adjacent teeth.
  * Normal vertical dimension with normal inter-arch space.

Exclusion Criteria:

* • Intra-bony lesions (e.g. cysts) or infections (e.g. abscess) that may retard the osteotomy healing.

  * General contraindications to implant surgery.
  * Subjected to irradiation in the head and neck area less than 1 year before implantation.
  * Untreated periodontitis.
  * Poor oral hygiene and motivation.
  * Uncontrolled diabetes.
  * Pregnant or nursing females.
  * Immunosuppressed or immunocompromised
  * Heavy smokers
  * Patients who undergo medication interfere with bone healing
  * Previous grafting procedures in the edentulous area.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Alveolar Ridge Horizontal Bone Gain | (CBCT) scans are taken preoperatively and 6 months postoperatively to evaluate bone changes. Superimposition of CBCT images is performed using Mimics 21.0 software (Materialise, Belgium) to assess bone augmentation
  measure the amount of horizontal bone gain achieved at the anterior mandibular ridge following horizontal ridge augmentation using either the computer-guided autogenous cortical shell technique or the free-hand technique.

SECONDARY OUTCOMES:
Accuracy of the Computer-assisted guide in the study group | Measured at: 6 months postoperatively using CBCT scans.
  CBCT superimposition is used to compare preoperative and postoperative ridge dimensions to determine how precisely the bone graft was placed.
  Measurement Tool: CBCT scans analyzed with Mimics 21.0 software
Intraoperative Time | During surgery by using a stopwatch.
  The total surgical duration for each technique is recorded to assess time efficiency.
  Measurement Tool: Stopwatch or surgical records. Unit of Measurement: Minutes.

IPD SHARING:
Plan to Share IPD: No